CLINICAL TRIAL: NCT05614401
Title: Long-term Efficacy of Remote Ischemic Postconditioning After Rt-PA Intravenous Thrombolysis in Patients With Acute Ischemic Stroke: The Randomized RESPONTH Trial
Brief Title: Long-term Outcome of RIPC After IV Thrombolysis in AIS Patients
Acronym: RESPONTH
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2022LSK-407
Record Dates: First submitted 2022-10-31; First posted 2022-11-14 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-10

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Functional Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RIPC group: Patients underwent RIPC treatment after IV thrombolysis in the index stroke.
  Interventions: Other: functional and medical information
- Control group: The control group underwent no inflations or deflations in the index stroke.
  Interventions: Other: functional and medical information

INTERVENTIONS:
Other: functional and medical information — 1) functional outcomes(mRS scoring), 2)survival status, 3) date of death in those who died (based on information of the treating physicians), 3) mRS score at the time of the interview, 4) recurrent stroke/TIA, 5) new onset atrial fibrillation, 6) other cardiovascular events, including myocardial infarction, pulmonary embolism, deep venous thrombosis, peripheral arteriopathy.

SUMMARY:
The goal of this observational study is to learn about the long-term efficacy of our previous study in acute ischemic stroke(AIS) patients who underwent either remote ischemic postconditioning(RIPC) or sham treatment after intravenous thrombolysis. The main questions it aims to answer are:

* Dose the RIPC treatment combined with IV thrombolysis can improve the long-term functional outcome in AIS patients?
* Dose the RIPC treatment combined with IV thrombolysis can improve the incidence rates of all-cause and cardiovascular mortality, recurrent stroke/TIA, new-onset clinical AF on this long-term follow-up? A single rater (A.E.P.) trained by an experienced stroke physician (S.T.E.) contacted patients, relatives, and family physicians to gather all available medical information on the following issues: 1) survival status, 2) date of death in those who died (based on information of the treating physicians), 3) mRS score at the time of the interview, 4) recurrent stroke/TIA, 5) new onset atrial fibrillation, 6) other cardiovascular events, including myocardial infarction, pulmonary embolism, deep venous thrombosis, peripheral arteriopathy.

Researchers will compare RIPC group and control group to see if the RIPC treatment have a long-term effect in AIS patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients who completed the previous interventional rater-blinded controlled study were invited for the follow-up session.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between August 2017 and June 2018, a total of 68 AIS patients who underwent IVT treatment were randomized into either the RIPC treatment group or the control group. During the trial period, thirty-four participants in the control group and thirty-two participants in the RIPC group were followed for the percentage of patients at 90 days with a favorable outcome, which was de- fined as a score of 0 or 1 on the modified Rankin Score (mRS). After the completion of the trial, the trial participants were followed by their primary care physicians.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
the proportion of excellent functional outcome, % | through study completion, an average of 5 year
  An excellent functional outcome define as mRS= 0 and 1.

SECONDARY OUTCOMES:
the proportion of favorable outcome (mRS scores 0-2), % | through study completion, an average of 5 year
  A favorable functional outcome define as mRS= 0-2.
incidence rates of all-cause and cardiovascular mortality, % | From date of randomization until the date of death from any cause, assessed up to 100 months
recurrent stroke/TIA | From date of randomization until the date of first documented recurrent stroke/TIA or date of death from any cause, whichever came first, assessed up to 100 months

CONTACTS AND LOCATIONS:
Overall Officials: Guoliang Li, Principal Investigator — First Affiliated Hospital of Xian Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiantong University, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] An J, Wei M, Wang D, Zhao C, Yuan X, Kimberly WT, Luo G, Li G. Long-term efficacy of remote ischaemic postconditioning after rt-PA intravenous thrombolysis in patients with acute ischaemic stroke. BMJ Open. 2025 Oct 28;15(10):e094001. doi: 10.1136/bmjopen-2024-094001. PMID 41151950